CLINICAL TRIAL: NCT05707559
Title: Knowledge Beliefs and Expectations of Chronic Musculoskeletal Patients About Their Physiotherapy Program
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, Principal Investigator, University of Thessaly
Other Study IDs: N8
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: chronic musculoskeletal pain; pain education; patient expectations; communication skills; physiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the knowledge, beliefs and expectations of patients with chronic musculoskeletal pain about their physiotherapy program and the relationship that they built with physiotherapists.

DETAILED DESCRIPTION:
The main questions of this study are:

Have patients with chronic pain educated in pain? To what extent physiotherapists use appropriate communication skills and show empathy? What expectations do the patients have of their rehabilitation program?

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic musculoskeletal pain more than 3 months and intensity more than 3/10 VAS.
* Greek speaking patients
* patients who are following or followed a physiotherapy treatment for their pain

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Musculoskeletal Patients
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | Baseline
  Questions will include participants' demographic characteristics (e.g. gender, age, education, employment status)
Knowledge about their pain | Baseline
  Fourteen questions about history of pain (e.g. intense, duration, area, other symptoms, radiation, previous history, diagnosis)
Pain (Neuroscience) Education | Baseline
  Patients will be asked whether they have received any education or explanation about their conditions from a healthcare professional (e.g. What have they learned about their pain? What do they know about pain neuroscience education? Whether it was explained to them and how understanding pain helped them?)
Patient's Experience about healthcare professional's communication skills | Baseline
  Seventeen questions on a five point Likert scale (1=never, 2= rarely, 3=sometimes, 4=often, 5=always). Questions adapted by the Calgary-Cambridge observation guide that delineates and structures the skills which aid doctor-patient communication.
Patient's Expectations | Baseline
  Four questions regarding patients' expectations for chronic pain management

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, PhD, Study Director — University of Thessaly
Locations (1):
- University of Thessaly, Lamia, Greece